CLINICAL TRIAL: NCT00983346
Title: Effect of Low Dose Bortezomib on Bone Formation in Smoldering Myeloma Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lab Staff that was required left the institution, therefore accrual closed prematurely
Sponsor: University of Utah (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HCI33979
Record Dates: First submitted 2009-09-22; First posted 2009-09-24 (Estimated); Results first posted 2015-11-30 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-07

CONDITIONS: Cancer; Myeloma; Multiple Myeloma
Keywords: cancer; myeloma; multiple myeloma; smoldering myeloma
MeSH Terms: conditions — Neoplasms; Neoplasms, Plasma Cell; Multiple Myeloma; Smoldering Multiple Myeloma | interventions — Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- All patients (Experimental): All participants enrolled.
  Interventions: Drug: Bortezomib

INTERVENTIONS:
Drug: Bortezomib — Bortezomib will be administered as a 3-5 second bolus IV injection at the dose of 0.7 mg/m2 on days 1, 8, 15, and 22 of each 42 day cycle.
  Patients will undergo nine 42-day cycles. At the end of this (day 378), patients will be assessed for bone remodeling changes. Evaluation for toxicities will be evaluated at the beginning of each cycle.
  Other Names: Velcade

SUMMARY:
OBJECTIVES

* Primary: To evaluate the bone anabolic effect of bortezomib in patients with smoldering myeloma.
* Secondary: To evaluate the effect of bortezomib on the natural history of smoldering myeloma.

DETAILED DESCRIPTION:
Smoldering multiple myeloma (SMM) is usually followed expectantly without therapy. The overall risk of progression to active multiple myeloma has been estimated up to 20% in the first year from diagnosis (Kyle et al, 2007). An angiogenic switch has been postulated as a pivotal event in the progression from MGUS to smoldering myeloma. Two trials for advanced and refractory MM patients tested this hypothesis using Thalidomide as antiangiogenic agent in association with biphosphonates showing and effect on disease progression (Barlogie et al, 2008).

The ubiquitin-proteasome pathway, which has been shown to be an essential cellular degradative system in myeloma cells, also regulates bone formation though effects on osteoblast differentiation (Pennisi et al., 2008).

Retrospective analysis of ALP variation in 2 large Bortezomib trials in the refractory setting confirmed the finding. In the SUMMIT trial (Zangari, et al., 2005), 77 patients were evaluated. The media increment ALP in levels of responding patients (patients with >50% decrease in paraprotein) upon completion of 3 cycles of therapy was statistically higher of those individuals with less than partial response (week 8, P=0.0015; responder range, 62-837 mL/L). In the APEX trial (Zangari et al. 2005), 422 patients were analyzed; 217 patients were randomized to bortezomib, 205 to dexamethasone. Within the bortezomib arm, the increment in serum ALP levels in responder patients (>CR) was statistically higher at week 3 (P=0.014), week 6 (P=0.002; responder rage, 31-272 mL/L) and week 9 (P=0.036). Comparing only responders patients in both arms of the study, we observed a significantly higher median ALP increase in the bortezomib compared to the dexamethasone arm (P<0.01; responder ran, 31-272 mL/L) (Zangari et al., 2007). A 25% increase in ALP (N=105) at week 6 was also the strongest indicator associated with quality of response (P<0.0001) and also with the time to progression (206 vs. 169 days) relative to patients with less than a 25% increase in ALP (N=228; P=0.01) (Zangari et al., 2007). We will now test the bone anabolic effect of bortezomib in a cohort of smoldering multiple myeloma patients.

Study rationale and selection of drug doses VELCADE has been shown to produce an anabolic bone effect (increase bone ALP and osteocalcin) in relapsed/refractory patients. This study will examine the bone anabolic effect in patients with smoldering myeloma who, with a median age of 67 years, have frequent evidence of osteopenia not associated with lytic bone disease. Risk of disease progression is estimated at 10% per year in this patient population. The primary aim of this trial is to determine the effect of a short course (i.e. 9 cycles) of low-dose Bortezomib on bone remodeling and on disease progression. The dose of bortezomib used in this trial of 0.7 mg/m2 is the lowest dose which has shown efficacy in the 3 largest monotherapy trials with bortezomib. Seventeen percent of patients in the APEX 9% of patients in CREST and 24% in SUMMIT trials were treated with 0.7 mg/m2 dosages. Bortezomib will be given on days 1, 8, 15, 22 over 42 days to reduce the incidence of possible drug related side effects.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosis of smoldering multiple myeloma
* Male or Female patients aged ≥ 18 years old
* Ability to provide written informed consent (obtained prior to participation in the study and any related procedures being performed) with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.
* Female subject is either post-menopausal or surgically sterilized or willing to use an acceptable method of birth control (i.e., a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) for the duration of the study
* Male subject agrees to use an acceptable method for contraception for the duration of the study.
* Serum M protein ≥3 g/dL and/or
* Bone marrow plasma cells ≥10%
* Absence of anemia, renal failure, hypercalcemia, and lytic bone lesions
* ANC ≥ 1.5 x 109 /L
* Hemoglobin ≥ 10g/dl
* Platelets ≥ 100 x 109 /L
* AST and ALT ≤2.5 x ULN
* Serum bilirubin ≤2.0 x ULN

Exclusion Criteria:

* Platelet count of <100 109/L within 14 days before enrollment.
* Absolute neutrophil count of <1.0 109/L within 14 days before enrollment.
* Creatinine clearance of <30 mL/minute within 14 days before enrollment.
* Patient has Grade 2 peripheral neuropathy within 14 days before enrollment.
* Myocardial infarction within 6 months prior to enrollment or has New York Heart Association (NYHA) Class III or IV heart failure (see section 8.4), uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Prior to study entry, any ECG abnormality at Screening has to be documented by the investigator as not medically relevant.
* Patient has hypersensitivity to bortezomib, boron or mannitol.
* Female subject is pregnant or breast-feeding. Confirmation that the subject is not pregnant must be established by a negative serum human chorionic gonadotropin (hCG) pregnancy test result obtained during screening. Pregnancy testing is not required for post-menopausal or surgically sterilized women.
* Patient has received other investigational drugs with 14 days before enrollment
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study.
* Diagnosed or treated for another malignancy within 3 years of enrollment, with the exception of complete resection of basal cell carcinoma or squamous cell carcinoma of the skin, an in situ malignancy, or low-risk prostate cancer after curative therapy.
* Patients currently taking bisphosphonates

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2009-10; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maurizio Zangari, MD, Principal Investigator — University of Utah
Locations (1):
- Huntsman Cancer Institute, Salt Lake City, Utah, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm -1 Bortezomib: All participants enrolled.
  Bortezomib: Bortezomib will be administered as a 3-5 second bolus IV injection at the dose of 0.7 mg/m^2 on days 1, 8, 15, and 22 of each 42 day cycle.
  Patients will undergo nine 42-day cycles. At the end of this (day 378), patients will be assessed for bone remodeling changes. Evaluation for toxicities will be evaluated at the beginning of each cycle.
Period: Overall Study
Arm/Group | Arm -1 Bortezomib
Started | 17
Completed | 17
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Arm -1 Bortezomib
Number analyzed (Participants) | 17
Age, Continuous [Median (Full Range); unit: years] | 61 [41 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 9

OUTCOME MEASURES:

1. Primary Outcome: Bone Anabolic Effect of Bortezomib in Patients With Smoldering Myeloma.
Description: The primary endpoint is the change in bone Alkaline Phosphatase at baseline and 6 weeks.
Time Frame: Baseline and 6 weeks
Population: Only 13 patents had bone alkaline phosphatase measured at the appropriate time points out of the 17 that completed the study
Measure: Number; unit: Percentage of Baseline Value
Groups:
- Arm 1 Bortezomib: All participants enrolled.
  Bortezomib: Bortezomib will be administered as a 3-5 second bolus IV injection at the dose of 0.7 mg/m2 on days 1, 8, 15, and 22 of each 42 day cycle.
  Patients will undergo nine 42-day cycles. At the end of this (day 378), patients will be assessed for bone remodeling changes. Evaluation for toxicities will be evaluated at the beginning of each cycle.
Arm/Group | Arm 1 Bortezomib
Number analyzed (Participants) | 13
Percentage of Baseline Value
  % Base Line Patient 1 | 178
  % Base Line Patient 3 | 105
  % Base Line Patient 4 | 105
  % Base Line Patient 6 | 99
  % Base Line Patient 7 | 95
  % Base Line Patient 8 | 119
  % Base Line Patient 10 | 128
  % Base Line Patient 11 | 84
  % Base Line Patient 13 | 125
  % Base Line Patient 14 | 120
  % Base Line Patient 15 | 96
  % Base Line Patient 16 | 98
  % Base Line Patient 17 | 431

ADVERSE EVENTS:
Arm/Group | Arm 1 Bortezomib
Serious Adverse Events (participants affected / at risk) | 2/17
Other Adverse Events (participants affected / at risk) | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 Bortezomib (N=17)
Obstruction of airway (Respiratory, thoracic and mediastinal disorders) | 1 (1)
back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
small bowel obstruction (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 Bortezomib (N=17)
abdomen pain (Gastrointestinal disorders) | 2 (2)
allergic reaction (Immune system disorders) | 1 (1)
altered mental status (Nervous system disorders) | 1 (2)
anxiety (Nervous system disorders) | 2 (2)
back pain (Musculoskeletal and connective tissue disorders) | 1 (3)
blurred vision (Eye disorders) | 1 (1)
bruising (Skin and subcutaneous tissue disorders) | 3 (3)
Candida albicans (Infections and infestations) | 1 (1)
cardiomegaly (Cardiac disorders) | 1 (1)
Chest pain (Musculoskeletal and connective tissue disorders) | 3 (3)
cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
depression (Nervous system disorders) | 1 (1)
diarrhea (Gastrointestinal disorders) | 1 (1)
dizziness (Nervous system disorders) | 2 (2)
dry eye syndrome (Eye disorders) | 1 (1)
ear discomfort (Ear and labyrinth disorders) | 1 (1)
edema (Blood and lymphatic system disorders) | 1 (1)
Elevated Ast (Metabolism and nutrition disorders) | 1 (1)
elevated Creatinine (Metabolism and nutrition disorders) | 3 (3)
elevated Prothrombin time (Blood and lymphatic system disorders) | 1 (1)
erythema (Skin and subcutaneous tissue disorders) | 1 (1)
falls (Injury, poisoning and procedural complications) | 1 (1)
fatigue (General disorders) | 7 (8)
finernail disocloration (General disorders) | 1 (1)
Headache (Nervous system disorders) | 3 (3)
Herpes lesion (Infections and infestations) | 1 (1)
Elevated LDL (Metabolism and nutrition disorders) | 1 (1)
Elevated VLDL (Metabolism and nutrition disorders) | 1 (1)
hyperbilirubinemia (Metabolism and nutrition disorders) | 2 (4)
hyperglycemia (Metabolism and nutrition disorders) | 4 (5)
hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
hypermagnesemia (Metabolism and nutrition disorders) | 1 (1)
hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (1)
hypoalbuminemia (Metabolism and nutrition disorders) | 2 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 6 (10)
Hypoesthesia (Nervous system disorders) | 1 (1)
hypokalemia (Metabolism and nutrition disorders) | 2 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 3 (3)
hypophoasphatemia (Metabolism and nutrition disorders) | 3 (9)
hypotension (Cardiac disorders) | 1 (1)
influenza (Infections and infestations) | 1 (1)
insomnia (Psychiatric disorders) | 3 (3)
Itching (Skin and subcutaneous tissue disorders) | 2 (2)
joint pain (Musculoskeletal and connective tissue disorders) | 2 (2)
leg pain (Musculoskeletal and connective tissue disorders) | 1 (1)
muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
nausea (Gastrointestinal disorders) | 2 (3)
neck ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1)
neuopathy (Nervous system disorders) | 5 (6)
night sweats (General disorders) | 1 (1)
nipple swelling (General disorders) | 1 (1)
Muscle pain (Musculoskeletal and connective tissue disorders) | 1 (1)
ovarian cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
elevated PSA (General disorders) | 1 (1)
Shoulder Pain (Musculoskeletal and connective tissue disorders) | 2 (2)
sinus congestion (Infections and infestations) | 1 (1)
skin redness (Skin and subcutaneous tissue disorders) | 1 (1)
sore throat (General disorders) | 1 (1)
Sublingual hematoma (Blood and lymphatic system disorders) | 1 (1)
sweating (General disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
tachycardia (Cardiac disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 5 (6)
toothache (General disorders) | 1 (1)
vomiting (Gastrointestinal disorders) | 1 (1)
Yersinia enterocolitica (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes